CLINICAL TRIAL: NCT07397416
Title: Intervention in the CPE Surveillance Algorithm and Isolation Re-evaluation With the Addition of PCR vs. Culture-based Protocol: Real-life Time Differences
Brief Title: Impact of Implementing a Rapid PCR-based Algorithm for Carbapenemase-producing Enterobacterales (CPE) and Infection Control Bundle in a Tertiary Hospital
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, EMILIO FELIPE HUAIER ARRIAZU, Emilio Felipe Huaier Arriazu, MD. Principal Investigator, Infection Control Committee, Hospital Italiano de Buenos Aires
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: CEPI No. 7443 PRIISA 15728
Record Dates: First submitted 2025-12-22; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Carbapenemase-Producing Enterobacterales (CPE) Colonization
Keywords: Healthcare-Associated Infections; Antimicrobial Resistance; Enterobacteriaceae Infections; Nosocomial Colonization; Infection Control
MeSH Terms: conditions — Cross Infection; Enterobacteriaceae Infections | interventions — Cytopathogenic Effect, Viral

STUDY DESIGN:
Intervention Model Description: This study follows a sequential, before-after interventional design. The same hospital population and inclusion criteria are applied in two consecutive periods:
  * Pre-intervention period: standard culture-based algorithm for carbapenemase-producing Enterobacterales (CPE) surveillance and isolation reevaluation.
  * Post-intervention period: implementation of a rapid PCR-based algorithm (BD MAX™ System) for CPE detection integrated into the same workflow.
  No randomization or masking is performed. The comparison evaluates real-life time differences in isolation and de-isolation processes before and after PCR implementation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-intervention period (No Intervention): The baseline phase preceding the implementation of the rapid PCR-based algorithm. During this period, the institutional workflow for carbapenemase-producing Enterobacterales (CPE) surveillance and isolation reevaluation relied exclusively on culture-based methods. Patients evaluated for CPE carriage or decolonization were tested using CHROMagar™ KPC and phenotypic confirmation methods (including MALDI-TOF and NG-Test CARBA 5 when indicated). Discontinuation of isolation required either three negative cultures or two negative cultures plus one PCR performed at least three months after the last positive result. No modification of staffing, alert systems, or isolation criteria occurred during this period.
- Post-intervention period (Active Comparator): The implementation phase beginning November 6, 2024, when the rapid PCR-based diagnostic algorithm for carbapenemase-producing Enterobacterales (CPE) was incorporated into the existing infection control workflow. Real-time PCR was performed using the BD MAX™ System to detect bla_KPC, bla_NDM, bla_VIM/IMP, and bla_OXA-48-like genes directly from rectal swabs. The infection control team coordinated sample requests, result communication, and isolation/de-isolation actions. The new algorithm prioritized PCR testing for surveillance and discontinuation of isolation in patients not receiving antibiotics, replacing culture-based testing in those scenarios.
  Interventions: Diagnostic Test: Rapid PCR-based algorithm for CPE detection

INTERVENTIONS:
Diagnostic Test: Rapid PCR-based algorithm for CPE detection — Implementation of a rapid real-time PCR-based diagnostic algorithm for the detection of carbapenemase-producing Enterobacterales (CPE) integrated into the institutional infection control workflow. The BD MAX™ System detects bla_KPC, bla_NDM, bla_VIM/IMP, and bla_OXA-48-like genes from rectal swabs. The infection control team manages the process from sample request to result-based isolation decision. The intervention began on November 6, 2024, upon availability of PCR supplies and reagents.
  Other Names: Rapid molecular diagnostic algorithm for CPE; BD MAX CPE PCR workflow
  Arms: Post-intervention period

SUMMARY:
Purpose:

Carbapenemase-producing Enterobacterales (CPE) are a growing cause of healthcare-associated infections, linked to high morbidity, mortality, and cost. Current screening methods rely mainly on culture, which can take up to 48 hours and delay infection control actions.

This study aims to evaluate the real-life impact of implementing a rapid PCR-based algorithm for CPE detection compared with the standard culture-based protocol, focusing on time differences in isolation and de-isolation decisions in hospitalized patients.

Design:

A quasi-experimental, before-and-after, retrospective study conducted at Hospital Italiano de Buenos Aires (HIBA).

Primary Outcome:

Time (in hours) between rectal swab request and change in isolation status (application or removal of isolation label) before and after PCR implementation.

Population:

Adult patients (≥18 years) admitted between October 2023-April 2024 (pre-intervention) and October 2024-April 2025 (post-intervention), who had contact isolation initiated or discontinued based on CPE surveillance results.

Rationale:

The introduction of rapid molecular testing could reduce operational delays and unnecessary isolation days, optimizing resource use in a setting with high CPE endemicity.

DETAILED DESCRIPTION:
Background:

Carbapenemase-producing Enterobacterales (CPE) are critical-priority pathogens associated with increased morbidity, mortality, and healthcare costs. Screening and isolation are recommended infection control measures, yet delays inherent to culture-based methods can hinder timely decision-making and overuse limited isolation rooms.

Objective:

To compare the time to initiation and discontinuation of contact isolation-from swab request to result availability and isolation status update-before and after implementing a rapid PCR-based diagnostic protocol for CPE identification.

Design and Setting:

Retrospective, quasi-experimental before-after study at the Hospital Italiano de Buenos Aires, Argentina. The pre-intervention period covers October 1, 2023-April 30, 2024; the post-intervention period covers October 1, 2024-April 30, 2025.

Intervention:

Incorporation of real-time PCR testing (BD MAX™ System) for CPE genes (bla_KPC, bla_NDM, bla_VIM/IMP, bla_OXA-48-like) into the existing CPE surveillance and isolation reevaluation workflow. The infection control team coordinates sample requests and response actions.

Primary Outcomes:

Time difference (in hours) from surveillance swab request to isolation implementation.

Time difference (in hours) from surveillance swab request to isolation discontinuation.

Secondary Outcomes:

Time differences stratified by weekday versus weekend.

Time differences according to sampling time (08:00-16:00 vs 16:00-08:00).

Time differences according to immunosuppression status.

Time differences in ICU versus general ward settings.

Data Collection:

Four timestamps will be extracted from the electronic health record (EHR): swab request, laboratory check-in, final laboratory result, and change in isolation logo. These will allow computation of operational intervals (request → action), collection delay, processing delay, and action delay.

Statistical Analysis:

Continuous variables will be summarized as medians and interquartile ranges. Median time differences between pre- and post-intervention periods will be compared using mixed-effects linear regression adjusted for immunosuppression, ICU admission, day of the week, and public holidays. Analyses will be conducted using Stata v16.

Ethical Considerations:

The study is retrospective and minimal-risk, involving only secondary use of clinical data. It has been submitted to the CEPI (Comité de Ética de Protocolos de Investigación), Hospital Italiano de Buenos Aires (PRIISA 15728), with waiver of informed consent under CIOMS 2019 Guideline 10.

Expected Impact:

By quantifying real-time process improvements after PCR implementation, this study will provide evidence on diagnostic turnaround times and operational efficiency in infection control practices.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged ≥18 years
* Patients screened for carbapenemase-producing Enterobacterales (CPE) carriage by perianal swab within the first 5 days of hospital admission
* Patients newly identified as CPE-colonized, leading to initiation of contact isolation
* Patients found to be decolonized, leading to discontinuation of contact isolation
* Patients with indication for active surveillance at hospital admission:

  * Transfer from another healthcare facility
  * Hospitalization in another healthcare center within the previous month
* Patients undergoing active surveillance during hospitalization:

  * First surveillance swab in high-risk neutropenic patients (HAR flag)
  * First surveillance swab in immunosuppressed units, such as hematopoietic stem-cell transplant wards
* Patients evaluated for discontinuation of contact precautions who meet all of the following:

  * Prior CPE-positive surveillance sample
  * At least 3 months since the last positive result and last hospitalization
  * No systemic antibiotic exposure during that period

Exclusion Criteria:

* Lost samples
* Insufficient samples
* Invalid laboratory test results requiring repeat sampling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Time from surveillance swab request to isolation implementation or discontinuation (hours) | From the date and time of electronic request for perianal swab collection until the date and time of isolation status update in the EHR, assessed up to 168 hours (7 days).
  Primary Outcome Measure
  1. Operational time from surveillance swab request to isolation status change (hours)
  Description:
  Time elapsed between the electronic request for perianal surveillance swab (clinical suspicion) and the implementation or discontinuation of the carbapenemase-producing Enterobacterales (EPC) isolation logo in the electronic health record (EHR).
  Unit of Measure: Hours

SECONDARY OUTCOMES:
Sample collection delay (hours) | From the date and time of electronic request for perianal swab collection until laboratory check-in of the sample, assessed up to 72 hours.
  Description:
  Time elapsed between the electronic request for perianal surveillance swab and laboratory check-in of the sample.
  Unit of Measure: Hours
Laboratory processing delay (hours) | From the date and time of laboratory check-in until the date and time of final laboratory result, assessed up to 96 hours.
  Time elapsed between laboratory check-in of the perianal swab sample and availability of the final laboratory result.
  Unit of Measure: Hours
Action delay after laboratory result (hours) | From the date and time of final laboratory result until the date and time of isolation status update in the EHR, assessed up to 72 hours.
  Time elapsed between availability of the final laboratory result and update of the EPC isolation status (logo) in the electronic health record.
  Unit of Measure: Hours

IPD SHARING:
Plan to Share IPD: No
Data derived from institutional electronic health records cannot be shared externally due to confidentiality agreements and national data protection laws (Law 25.326, Argentina). Aggregated results will be available upon publication.

REFERENCES:
- [Result] al-Hasany M, Mohamed AS. Veno-occlusive disease of the liver in Iraq. Nine cases occurring in three Bedouin families. Arch Dis Child. 1970 Oct;45(243):722-4. doi: 10.1136/adc.45.243.722. No abstract available. PMID 5477705
- [Result] Kinasewitz GT, Welch MH. A simple method to assess postoperative risk. Chest. 2001 Oct;120(4):1057-8. doi: 10.1378/chest.120.4.1057. No abstract available. PMID 11591537
- [Result] Ruszymah BH, Nabishah BM, Aminuddin S, Khalid BA. Effects of glycyrrhizic acid on right atrial pressure and pulmonary vasculature in rats. Clin Exp Hypertens. 1995 Apr;17(3):575-91. doi: 10.3109/10641969509037425. PMID 7613529
- [Result] Posey BL, Kimble SN. Quantitative determination of 11-nor-delta 9-tetrahydrocannabinol-9-carboxylic acid in urine by HPLC. J Anal Toxicol. 1984 Sep-Oct;8(5):234-8. doi: 10.1093/jat/8.5.234. PMID 6094916
- [Result] A C, N C, A S, A P, E Y, F G, M C. Validation of a rapid molecular detection test for gram-negative multidrug-resistant bacteria in rectal swabs upon admission of patients to the intensive care unit. Diagn Microbiol Infect Dis. 2024 Jun;109(2):116250. doi: 10.1016/j.diagmicrobio.2024.116250. Epub 2024 Mar 8. PMID 38479092
- [Result] Fasciana T, Antonelli A, Bianco G, Lombardo D, Codda G, Roscetto E, Perez M, Lipari D, Arrigo I, Galia E, Tricoli MR, Calvo M, Niccolai C, Morecchiato F, Errico G, Stefani S, Cavallo R, Marchese A, Catania MR, Ambretti S, Rossolini GM, Pantosti A, Palamara AT, Sabbatucci M, Serra N, Giammanco A. [The CCM Project "Phenotypic and molecular screening methodologies for the detection of coloniza-tions due to carbapenem-resistant Enterobacterales (CRE)"]. Epidemiol Prev. 2024 Nov-Dec;48(6):470-475. doi: 10.19191/EP24.6.A806.137. Italian. PMID 39679488
- [Result] Lydeamore MJ, Wu D, Donker T, Gorrie C, Higgs CK, Easton M, Hennessy D, Geard N, Howden BP, Cooper BS, Wilson A, Peleg AY, Stewardson AJ. Changes in isolation guidelines for CPE patients results in only mild reduction in required hospital beds. Infect Dis Health. 2025 May;30(2):128-131. doi: 10.1016/j.idh.2024.10.004. Epub 2024 Nov 24. PMID 39586760
- [Result] Jimenez A, Fennie K, Munoz-Price LS, Ibrahimou B, Pekovic V, Abbo LM, Martinez O, Rosello G, Sposato K, Doi Y, Trepka MJ. Duration of carbapenemase-producing Enterobacteriales carriage among ICU patients in Miami, FL: A retrospective cohort study. Am J Infect Control. 2021 Oct;49(10):1281-1286. doi: 10.1016/j.ajic.2021.06.006. Epub 2021 Jun 17. PMID 34146625
- [Result] Zimmerman FS, Assous MV, Bdolah-Abram T, Lachish T, Yinnon AM, Wiener-Well Y. Duration of carriage of carbapenem-resistant Enterobacteriaceae following hospital discharge. Am J Infect Control. 2013 Mar;41(3):190-4. doi: 10.1016/j.ajic.2012.09.020. PMID 23449280
- [Result] van Veen A, de Goeij I, Damen M, Huijskens EGW, Paltansing S, van Rijn M, Bentvelsen RG, Veenemans J, van der Linden M, Vos MC, Severin JA; Infection Prevention and Antimicrobial Resistance Care Network South-western Netherlands. Regional variation in the interpretation of contact precautions for multi-drug-resistant Gram-negative bacteria: a cross-sectional survey. J Hosp Infect. 2024 Oct;152:1-12. doi: 10.1016/j.jhin.2024.06.020. Epub 2024 Jul 26. PMID 39069006
- See also: Surveillance of antimicrobial resistance in Europe 2017. In: European Centre for Disease Prevention and Control — https://www.ecdc.europa.eu/en/publications-data/surveillance-antimicrobial-resistance-europe-2017
- See also: Prevention I. Guidelines for the prevention and control of carbapenem-resistant Enterobacteriaceae, Acinetobacter baumannii and Pseudomonas aeruginosa in health care facilities. World Health Organization; 1 Nov 2017 — https://www.who.int/publications/i/item/guidelines-for-the-prevention-and-control-of-carbapenem-resistant-enterobacteriaceae-acinetobacter-baumannii-and-pseudomonas-aeruginosa-in-health-care-facilities
- See also: Nov. ALGORITMOS DE DETECCIÓN DE CARBAPENEMASAS 2024. — http://antimicrobianos.com.ar/2024/11/algoritmos-de-deteccion-de-carbapenemasas-2024/